CLINICAL TRIAL: NCT00949806
Title: Phase II Non Comparative, Open Study to Assess the Efficacy and Safety of the Botulinum Toxin Type A in Patients With Restless Legs Syndrome (RLS)
Brief Title: Restless Legs Syndrome Treatment With Botulinum Toxin
Acronym: SOXIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: IPSEN PHARMA S.A.S (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2008/35
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Restless Legs Syndrome
Keywords: Botulinum toxin
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Injections, Intradermal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Administrated (Experimental): All patients included will receive an intradermal administration of BNT
  Interventions: Drug: BNT (intradermal injection)

INTERVENTIONS:
Drug: BNT (intradermal injection) — Patients with severe RLS will receive a one-time intradermal administration of BNT into the most symptomatic areas of both legs.
  Injections will be distributed in a grid distribution pattern covering a total of 20 equidistant sites per symptomatic area. Each symptomatic area will receive a maximum 250 units of BNT (12.5 units per injection). The total BNT injected units should not exceed 1000 units per patient.

SUMMARY:
Restless Legs Syndrome (RLS) is a common sensori-motor disorder that causes sensory discomfort and motor restlessness, most often in the legs, which improves with movement. Although medications are available to treat the disorder, many people either experience side effects that prevent them from continuing on the medication or do not sufficiently respond to current RLS medications. Recently, botulinum toxin type A (BNT) has been reported to relief RLS in patients with severe symptoms but this was not confirmed by other anecdotal reports. The investigators propose to test the efficacy of BNT on RLS symptoms by designing a more controlled study. Ultimately, this may lead to extend the therapeutic arsenal of this disorder.

DETAILED DESCRIPTION:
The restless legs syndrome (RLS) is a chronic sensori-motor disorder affecting an estimated 7.2% to 11.5% of the adult population. It is characterised by a complaint of an irresistible urge to move the legs. This urge can often be accompanied by pain or other uncomfortable and unpleasant sensations, it either occurs or worsens with rest particularly at night, and improves with activity. RLS is diagnosed clinically by means of the four essential criteria established by the International Restless Legs Syndrome Study Group.

There is still no comprehensive understanding of the underlying pathophysiological processes of RLS, but the evidence for a primary dopaminergic role in RLS is to be found in the excellent pharmacological response to low-dose dopaminergic medications. Another recent evidence suggests an enhanced sensitization of central pain processing in patients with RLS. This had led to consider the botulinum toxin type A (BNT) as an alternative treatment in patients refractory to current RLS medications or in those suffering from adverse events. The therapeutic benefit of BNT injection in patients with recalcitrant RLS has been anecdotally reported lately but not confirmed by other reports.

The aim of our study is to evaluate the efficacy and tolerance of intradermal BNT injection in severely affected patients with idiopathic RLS.

For this we designed a phase II non comparative, open study. Patients with severe RLS will receive a one-time intradermal administration of BNT into the most symptomatic areas of both legs. Injections will be distributed in a grid distribution pattern covering a total of 20 equidistant sites per symptomatic area. Each symptomatic area will receive a maximum 250 units of BNT (12.5 units per injection). The total BNT injected units should not exceed 1000 units per patient.

Outcome measures will be evaluated at baseline, then at 2, 6, 12, 18 and 24 weeks following BNT administration and assessed by mean of the International RLS Rating Scale and Clinical Global Impression Scale.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 years old
* Normal neurological clinical examination
* A minimum score of 21 on the RLS severity rating scale
* Primary RLS diagnosis based on (i) the presence of a characteristic clinical history and on (ii) the International Restless Legs Syndrome Study Group (IRLSSG) diagnostic criteria.
* Medications regimen for RLS must be stabilized for more than 6 weeks prior to entering the study
* informed consent

Exclusion Criteria:

* Medical history of diabetes, depression, kidney failure, myasthenia
* Iron deficiency
* Pregnancy, lactation, woman of childbearing age without efficient contraceptive method
* Patient undergoing aminosid antibiotherapy or BNT injection for other indication
* Any contra-indication to BNT injection
* Participation to other clinical study within 30 days
* Patient under any administrative or legal supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of BNT in the treatment of RLS measured by at least 50% improvement of the RLS severity score as measured by the International Restless Legs Syndrome Severity Scale (IRLSRS) at day 15 following BNT injection | Outcome measures will be evaluated at baseline, then at 2, 6, 12, 18 and 24 weeks.

SECONDARY OUTCOMES:
Efficacy duration (maintenance of at least 50% improvement of the RLS severity on the IRLSRS at week 6, 12, 18 and 24 compared to baseline severity score | Outcome measures will be evaluated at baseline, then at 2, 6, 12, 18 and 24 weeks
Adverse events of BNT injection | Outcome measures will be evaluated at baseline, then at 2, 6, 12, 18 and 24 weeks
Clinical Global Impression (CGI) improvement | Outcome measures will be evaluated at baseline, then at 2, 6, 12, 18 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Imad GHORAYEB, MD, PhD, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- CHU de Bordeaux, Pessac, France

REFERENCES:
- [Background] Rotenberg JS, Canard K, Difazio M. Successful treatment of recalcitrant restless legs syndrome with botulinum toxin type-A. J Clin Sleep Med. 2006 Jul 15;2(3):275-8. PMID 17561538
- [Background] Ghorayeb I, Burbaud P. Failure of botulinum toxin A to relieve restless legs syndrome. Sleep Med. 2009 Mar;10(3):394-5. doi: 10.1016/j.sleep.2008.03.002. Epub 2008 May 29. No abstract available. PMID 18514023
- [Background] Nahab FB, Peckham EL, Hallett M. Double-blind, placebo-controlled, pilot trial of botulinum toxin A in restless legs syndrome. Neurology. 2008 Sep 16;71(12):950-1. doi: 10.1212/01.wnl.0000325994.93782.a1. No abstract available. PMID 18794499
- [Derived] Ghorayeb I, Benard A, Vivot A, Tison F, Burbaud P. A phase II, open-label, non-comparative study of Botulinum toxin in Restless Legs Syndrome. Sleep Med. 2012 Dec;13(10):1313-6. doi: 10.1016/j.sleep.2012.08.019. Epub 2012 Oct 11. PMID 23063302